CLINICAL TRIAL: NCT03615495
Title: Flourish Pediatric Esophageal Atresia Device Post-Approval Study (Flourish)
Brief Title: Flourish™ Pediatric Esophageal Atresia
Status: Completed | Type: Observational
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Other Study IDs: 17-09
Record Dates: First submitted 2018-07-31; First posted 2018-08-03 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Esophageal Atresia; Digestive System Abnormalities; Esophageal Disorders Congenital
Keywords: Esophageal; Atresia; Congential
MeSH Terms: conditions — Esophageal Atresia; Digestive System Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Flourish device: The Flourish Pediatric Esophageal Atresia device is indicated for use in lengthening atretic esophageal ends and creating an anastomosis with a non-surgical procedure in pediatric patients.
  Interventions: Device: Flourish Pediatric Esphogeal Atresia device

INTERVENTIONS:
Device: Flourish Pediatric Esphogeal Atresia device — The Flourish Pediatric Esophageal Atresia device consists of an esophageal catheter and a gastric catheter. Both catheters are equipped with an inner magnet catheter. When the esophageal and gastric catheters are aligned tip to tip, the magnets attract.

SUMMARY:
This study is continued evaluation of the safety and probable benefit of the Flourish Pediatric Esophageal Atresia device through the Humanitarian Device Exemption (HDE) pathway.

ELIGIBILITY:
Inclusion Criterion:

* Patient treated for esophageal atresia with Flourish device starting May 12, 2017

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with esophageal atresia without a tracheoesophageal fistula (TEF) or for whom a concurrent TEF has been closed as a result of a prior procedure.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Rate of Adverse Events | 2 years
  Adverse Events include: stricture at the anastomotic site leading to the need for dilation or surgery and peri-anastomotic leaks

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - Hawaii, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Brenner Children's Hospital, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center, Dallas, Texas
  - Carilion Children's Hospital, Roanoke, Virginia
  - American Family Children's Hospital, Madison, Wisconsin
- McGill University Department of Pediatric Surgery, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Cook Research Incorporated (CRI) is fully committed to supporting the principles of responsible data sharing, including providing qualified scientific researchers access to deidentified, patient-level data from CRI clinical studies to conduct legitimate scientific research. Data underlying the results reported in this clinical study will be made available for request immediately after approval or clearance of the product and ending 5 years after approval or clearance. Interested researchers may review the "Cook Research Incorporated Policy on Access to Clinical Study Data" at https://www.cookresearchinc.com/extranet/data-access.html and submit a complete research proposal to request data access. Additional study documents (such as the study protocol) will be shared as needed if the data access request is granted. A data sharing agreement will be executed for access to deidentified patient-level data.